CLINICAL TRIAL: NCT04981093
Title: Effect of Dexamethasone on Postoperative Inflammatory Factors in Elderly Patients Undergoing Lunmbar Spine Surgery
Brief Title: Effect of Dexamethasone on Postoperative Inflammatory Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2020-519
Record Dates: First submitted 2021-06-14; First posted 2021-07-28 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2021-07

CONDITIONS: Inflammation
Keywords: intravenous dexamethasone; inflammation; QoR15; drainage
MeSH Terms: conditions — Inflammation | interventions — Calcium Dobesilate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Dexamethasone (Experimental): Group dexamethasone patients received intravenous injection after anesthesia induction
  Injection 0.15mg/kg dexamethasone (2ml）
  Interventions: Drug: Dexamethasone Injection
- Group Saline (Placebo Comparator): Group Control patients were also given 2ml of normal saline intravenously after induction of anesthesia
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexamethasone Injection — Intravenous injection after induction of anesthesia
  Injection 0.15mg/kg dexamethasone (2ml)
  Arms: Group Dexamethasone
Drug: Normal saline — 2ml of normal saline was injected intravenously after induction of anesthesia
  Arms: Group Saline

SUMMARY:
This topic foe randomized prospective study.Detection of elderly patients with lunmbar spinal postoperative inflammatory substances in the blood and drainage of liquid level ,clear whether low-dose dexamethasone can inhibit the inflammation, the observation of elderly patients with lumbar spinal postoperative drainage star, to explor whether low-dose dexamthasone can reduce postoperative incision drainage, thus impove the postoprative drainage tube pull rate within three days, which in turn reduce because of the place a retrograde infection caused by drainage tube.

DETAILED DESCRIPTION:
A total of 100 patients undergoing posterior lumbar disc fusion were randomly divided into control group (group C,n=50) and dexamethasone group (group D,n=50). Group D was given 0.15mg/kg dexamethasone (2ml) intravenously after anesthesia induction. Group C was also intravenously injected with 2ml normal saline after anesthesia induction.On this basis, monitor the main results and secondary results

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥65years of age
* American Society of Anesthesiologists (ASA) physical status 2-4
* Elective or expedited non-cardiac surgery of at least 2 hours dura- tion under general anaesthesia
* Requiring a hospital stay of at least one postoperative night
* A surgical skin incision >5 cm in length or multiple incisions with a total incision length of >5 cm

Exclusion Criteria:·

* Poorly controlled diabetes (HbA1c>9.0%)
* Endovascular procedure with a small (<5 cm length) skin incision Ophthalmic surgery
* Planned dexamethasone (or other corticosteroid) therapy (eg, history of intractable PONV, maxillofacial surgery, intracranial neurosurgery)
* Recent (<2 weeks since end of treatment) infective episode requir- ing treatment with antibiotics
* Chronic antibiotic therapy (eg, for bronchiectasis, cystic fibrosis etc)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
the change of drainage fluid volume | 6 hours after surgery， the morning of 1, 2, and 3 days after surgery
  Drainage fluid （ml）was collected and the volume of drainage fluid was recorded
  Until the drainage tube was pulled out,
the change of Inflammatory mediators in the drainage fluid | 6 hours after surgery， the morning of 1, 2, and 3 days after surgery
  CRP(mg/ L) in postoperative drainage fluid was observed

SECONDARY OUTCOMES:
the change of blood inflammatory mediators | 6 hours after surgery， the morning of 1, 2, and 3 days after surgery
  Fasting blood was collected from each enrolled patient preoperatively, 6 hours after surgery and on the morning of 1, 2, and 3 days after surgery
  Fasting blood, blood samples were centrifuged (1500r/min, 15min) and serum was separated and placed in -80℃ deep low temperature refrigerator for measurement. The observation technique
  After the blood CRP(mg/l)
the change of blood routine white blood cell count | 6 hours after surgery， the morning of 1, 2, and 3 days after surgery
  Fasting blood was collected from each enrolled patient preoperatively, 6 hours after surgery and on the morning of 1, 2, and 3 days after surgery
  Fasting blood, blood samples were centrifuged (1500r/min, 15min) and serum was separated and placed in -80℃ deep low temperature refrigerator for measurement. The observation technique
  After the blood blood routine white blood cell count

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corcoran TB, Myles PS, Forbes AB, O'Loughlin E, Leslie K, Story D, Short TG, Chan MT, Coutts P, Sidhu J, Cheng AC, Bach LA, Ho KM; Australian and New Zealand College of Anaesthetists Clinical Trials Network (ANZCA), and the Australian Society for Infectious Diseases (ASID) Clinical Research Network. The perioperative administration of dexamethasone and infection (PADDI) trial protocol: rationale and design of a pragmatic multicentre non-inferiority study. BMJ Open. 2019 Sep 6;9(9):e030402. doi: 10.1136/bmjopen-2019-030402. PMID 31494615
- [Background] Corcoran TB, Myles PS, Forbes AB, Cheng AC, Bach LA, O'Loughlin E, Leslie K, Chan MTV, Story D, Short TG, Martin C, Coutts P, Ho KM; PADDI Investigators; Australian and New Zealand College of Anaesthetists Clinical Trials Network; Australasian Society for Infectious Diseases Clinical Research Network. Dexamethasone and Surgical-Site Infection. N Engl J Med. 2021 May 6;384(18):1731-1741. doi: 10.1056/NEJMoa2028982. PMID 33951362